CLINICAL TRIAL: NCT05389774
Title: DOLCE: Determining the Impact of Optellum's Lung Cancer Prediction (LCP) Artificial Intelligence Solution on Service Utilisation, Health Economics and Patient Outcomes
Brief Title: DOLCE: Determining the Impact of Optellum's Lung Cancer Prediction Solution
Acronym: DOLCE
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Optellum Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21RM052
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: AI (Artificial Intelligence); Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple; Lung Cancer
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-centre prospective observational cohort study recruiting patients with 5-30mm solid and part-solid pulmonary nodules that have been detected on CT chest scans performed as part of routine practice. The aim is to determine whether physician decision making with the AI-based LCP tool, generates clinical and health-economic benefits over the current standard of care of these patients.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all of the following apply:

* Are aged 35 years or above
* Have baseline CT study with at least one incidentally detected solid or part-solid (must have a solid component >=80%) pulmonary nodule that:

  * is not fully calcified
  * Is 5-30mm inclusive in maximum axial diameter for the whole lesion measured using manual electronic callipers
* Have baseline CT study that includes at least one series that meets all of the following (training for this will be provided):

  * Is of a type that meets VNC instructions for use
  * Comprises at least one full-inspiration breath-hold scans without a high degree of contrast media and does not exhibit quality issues (e.g., motion artefacts)

Exclusion Criteria:

Patients will be excluded from the study if any of the following apply:

* Have received a diagnosis for cancer in the last 5 years
* Have thoracic implants that impact the image appearance of the nodule
* Have more than five reported pulmonary nodules of any size or type excluding fully calcified nodules (this criterion is used as a proxy due to the risk of being an infection or metastasis)
* Have one or more additional nodules where any of the following applies:

  * Are already undergoing follow-up according to pulmonary nodule management standard care
  * Pure ground glass opacity (GGO) of >=5mm in maximum axial diameter for the whole lesion measured using manual electronic callipers
  * >30mm in maximum axial diameter for the whole lesion measured using manual electronic callipers

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CT scans of patients for whom a pulmonary nodule has been identified will be reviewed for study eligibility by a member of the local site's clinical team for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Determine the potential effect of the LCP on discharge | up to 1 year.
  Measured difference between standard care, LCP and LCP-guided care for:
  * Percentage of cancer patients discharged (straight after assessment of the baseline scan)
  * Percentage of benign-nodule patients discharged (straight after assessment of the baseline scan)

SECONDARY OUTCOMES:
Determine the potential effect of the LCP on overall clinical management, as well as scan and procedure utilization. | up to 1 year.
  Percentage of cancer patients for whom there would have been a change in clinical management by LCP and LCP-guided care compared with the actual (standard) care (correctly by more aggressive management and incorrectly for less aggressive management).
  Percentage of benign-nodule patients for whom there would have been a change in clinical management by LCP and LCP-guided care compared with the actual (standard) care (incorrectly by more aggressive management and correctly for less aggressive management).
  Measured difference between standard care, LCP and LCP-guided care for:
  * Percentage of CT scans and PET/CT scans performed on benign-nodule patients
  * Percentage of non-surgical biopsies performed on benign-nodule patients
  * Percentage of surgical excisions on benign-nodule patients
Determine the potential effect of the hypothetical LCP-informed care versus standard care on patient outcomes. | up to 1 year.
  Measured difference between standard care, LCP and LCP-guided care for:
  * Percentage of thoracic, respiratory or vascular events related to biopsies or surgical excisions for lung nodules or suspected lung cancer occurring within 30 days of the procedure on benign-nodule patients
  * Percentage of lung cancers stratified by stage
  * Time in days between nodule detection and lung cancer diagnosis
Determine the potential health-economic effect of the hypothetical LCP-informed care versus standard care | up to 1 year.
  Measured difference between standard care, LCP and LCP-guided care for:
  * The composite standardized GBP costs of all healthcare-related activity for lung nodules or suspected lung cancer
  * Health-related utilities (life years and QALYs)
Determine the potential effect of the LCP on possible adherence to clinical guidelines. | up to 1 year.
  Measured difference between standard care and LCP-guided care for :
  Number and percentage of patients for whom a validated risk model (Brock or LCP) is used to guide the next clinical management step (i.e., counting the instances where Brock is not used, or where LCP is not possible to compute or it is ignored).

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Betsi Cadwaladr University Health Board, Bangor
  - Frimley Health NHS Foundation Trust (Wexham Park Hospital), Frimley
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - King's College Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - St. George's University Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

REFERENCES:
- [Derived] O'Dowd E, Berovic M, Callister M, Chalitsios CV, Chopra D, Das I, Draper A, Garner JL, Gleeson F, Janes S, Kennedy M, Lee R, Mauri F, McKeever TM, McNulty W, Murray J, Nair A, Park J, Rawlinson J, Sagoo GS, Scarsbrook A, Shah P, Sudhir R, Talwar A, Thakrar R, Watkins J, Baldwin DR. Determining the impact of an artificial intelligence tool on the management of pulmonary nodules detected incidentally on CT (DOLCE) study protocol: a prospective, non-interventional multicentre UK study. BMJ Open. 2024 Jan 4;14(1):e077747. doi: 10.1136/bmjopen-2023-077747. PMID 38176863